CLINICAL TRIAL: NCT04440176
Title: A PHASE 2b, RANDOMIZED, OBSERVER-BLINDED TRIAL TO DESCRIBE THE SAFETY, TOLERABILITY, AND IMMUNOGENICITY OF MenABCWY ADMINISTERED ON 2 DIFFERENT DOSING SCHEDULES IN HEALTHY PARTICIPANTS ≥11 TO <15 YEARS OF AGE
Brief Title: A Trial to Describe the Safety and Immunogenicity of MenABCWY When Administered on 2 Schedules
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: C3511004; 2019-004923-19 (EudraCT Number)
Record Dates: First submitted 2020-06-15; First posted 2020-06-19 (Actual); Results first posted 2025-01-08 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2024-12

CONDITIONS: Meningococcal Vaccine
Keywords: pentavalent meningococcal vaccine
MeSH Terms: interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group 1 (MenABCWY 0-, 12-months) (Experimental): MenABCWY administered at Month 0 and Month 12
  Interventions: Biological: MenABCWY
- Group 2 (MenABCWY 0-, 36-months) (Experimental): MenABCWY administered at Month 0 and Month 36
  Interventions: Biological: MenABCWY; Biological: Saline

INTERVENTIONS:
Biological: MenABCWY — Neisseria meningitidis group A, B, C, W, and Y vaccine
  Other Names: pentavalent meningococcal vaccine
Biological: Saline — Placebo
  Arms: Group 2 (MenABCWY 0-, 36-months)

SUMMARY:
This study is designed to describe the short-term immunogenicity and safety of 2 doses of Neisseria meningitidis group A, B, C, W, and Y vaccine (MenABCWY) separated by either 12 or 36 months during adolescence, and immunopersistence up to 24 months after completing 2 doses separated by a 12-month interval.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants 11 through <15 years of age at the time of randomization.
* Participants who have never received a prior dose of any meningococcal vaccine. Written confirmation of vaccination history must be obtained prior to randomization.
* Available for the entire study period and can be reached by telephone.
* Healthy participant as determined by medical history, physical examination, and judgement of the investigator.
* Negative urine pregnancy test for all female participants; pregnancy test is not applicable to male participants.

Exclusion Criteria:

* A previous anaphylactic reaction to any vaccine or vaccine-related component.
* Bleeding diathesis or condition associated with prolonged bleeding time that would contraindicate intramuscular injection.
* A known or suspected defect of the immune system that would prevent an immune response to the vaccine, such as participants with congenital or acquired defects in B-cell function, those receiving chronic systemic (oral, intravenous, or intramuscular) corticosteroid therapy, or those receiving immunosuppressive therapy.
* History of microbiologically proven disease caused by Neisseria meningitidis or Neisseria gonorrhoeae.
* Significant neurological disorder or history of seizure (excluding simple febrile seizure).
* Any neuroinflammatory or autoimmune condition, including, but no limited to, transverse myelitis, uveitis, optic neuritis, and multiple sclerosis.
* Participants receiving any allergen immunotherapy with a nonlicensed product or receiving allergen immunotherapy with a licensed product and are not on stable maintenance doses.
* Receipt of any blood products, including immunoglobulin, within 6 months before the first study vaccination.
* Current use of systemic antibiotics with no foreseeable date of discontinuation prior to anticipated date of enrollment (first vaccination).

Ages: 11 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 309 (Actual)
Dates: Start 2020-06-17 (Actual); Primary Completion 2024-01-05 (Actual); Study Completion 2024-01-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (19):
- United States (19):
  - Alliance for Multispecialty Research, LLC, Mobile, Alabama
  - California Research Foundation, San Diego, California
  - Nona Pediatric Center, Orlando, Florida
  - Velocity Clinical Research, Norfolk, Norfolk, Nebraska
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Ohio Pediatric Research Association Inc., Dayton, Ohio
  - Coastal Carolina Research Center, North Charleston, South Carolina
  - Benchmark Research, Fort Worth, Texas
  - Texas Health Resources, Fort Worth, Texas
  - Diagnostics Research Group, San Antonio, Texas
  - Wee Care Pediatrics, Kaysville, Utah
  - Wasatch Pediatrics, Cottonwood Office, Murray, Utah
  - Utah Valley Pediatrics - Timpanogos Office, Orem, Utah
  - Alliance for Multispecialty Research, LLC, Roy, Utah
  - J. Lewis Research, Inc. / Foothill Family Clinic, Salt Lake City, Utah
  - J. Lewis Research, Inc. / Foothill Family Clinic South, Salt Lake City, Utah
  - Alliance for Multispecialty Research, LLC, South Jordan, Utah
  - Wee Care Pediatrics, Syracuse, Utah
  - Pediatric Research of Charlottesville, LLC, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C3511004

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 309 participants were enrolled and randomized to receive study vaccination in this study out of which, 300 participants were vaccinated.
Pre-assignment Details: Participants aged greater than or equal to (>=) 11 years to less than (<) 15 years were randomized to receive Neisseria meningitidis Group A, B, C, W, and Y (MenABCWY) vaccine either at 0-and 12-Month schedule (Group 1) or at 0- and 36-Month schedule (Group 2).
Groups:
- Group 1 (MenABCWY 0- and 12-Month Schedule): Participants were randomized to receive 0.5 milliliter (mL) of MenABCWY vaccine intramuscularly on Day 1/Month 0 (Vaccination 1) and at Month 12 (Vaccination 2).
- Group 2 (MenABCWY 0- and 36-Month Schedule): Participants were randomized to receive 0.5 mL of MenABCWY vaccine intramuscularly on Day 1/Month 0 (Vaccination 1), and at Month 36 (Vaccination 3). Participants received 0.5 mL of placebo (normal saline) intramuscularly at Month 12 (Vaccination 2).
Period: Overall Study
Arm/Group | Group 1 (MenABCWY 0- and 12-Month Schedule) | Group 2 (MenABCWY 0- and 36-Month Schedule)
Started | 155 | 154
Safety Population (Received at least 1 dose of vaccine and had safety data post vaccination) | 146 | 148
Completed | 102 | 102
Not Completed | 53 | 52
Not completed — Withdrawal by Subject | 5 | 3
Not completed — Withdrawal by parent/guardian | 4 | 5
Not completed — Adverse Event | 2 | 6
Not completed — Lost to Follow-up | 22 | 23
Not completed — Medication error without associated adverse event | 0 | 1
Not completed — No longer met eligibility criteria | 7 | 1
Not completed — Other | 1 | 2
Not completed — Protocol deviation | 6 | 8
Not completed — Randomized but not vaccinated | 6 | 3

BASELINE CHARACTERISTICS:
Population: Safety population set included all randomized participants who received at least 1 dose of the study intervention and had safety data reported after vaccination. As per statistical analysis plan safety population was used to for baseline characteristics evaluation.
Groups:
- Group 1 (MenABCWY 0- and 12-Month Schedule): Participants were randomized to receive 0.5 mL of MenABCWY vaccine intramuscularly on Day 1/Month 0 (Vaccination 1) and at Month 12 (Vaccination 2).
- Total: Total of all reporting groups
Arm/Group | Group 1 (MenABCWY 0- and 12-Month Schedule) | Group 2 (MenABCWY 0- and 36-Month Schedule) | Total
Number analyzed (Participants) | 146 | 148 | 294
Age, Continuous [Mean (Standard Deviation); unit: Years] | 11.5 (0.65) | 11.5 (0.65) | 11.5 (0.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65 | 66 | 131
  Male | 81 | 82 | 163
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 22 | 32 | 54
  Not Hispanic or Latino | 123 | 116 | 239
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 3 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 10 | 14 | 24
  White | 125 | 126 | 251
  More than one race | 5 | 5 | 10
  Unknown or Not Reported | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Serum Bactericidal Assay Using Human Complement (hSBA) Titer >=Lower Limit of Quantitation (LLOQ) for Each of the 4 Primary Neisseria Meningitidis Serogroup B (MenB) Test Strains at Baseline: 0 and 12 Month Schedule
Description: Percentage of participants achieving hSBA titer >=LLOQ (1:16 for strain A22 and 1:8 for strains A56, B24, and B44) for each of the 4 primary MenB test strains at baseline were reported in this outcome measure. Here, 'Post Vaccination 2 Evaluable Population'=PV2 EP and "Number analyzed" = number of participants evaluable at specific rows.
Time Frame: Baseline (before vaccination 1)
Population: PV2 EP : all randomized participants, eligible throughout 1 month after second dose of MenABCWY; received vaccine at visit(V)1 for groups(G) 1 and 2,V4 for G1, V9 for G2;blood drawn for assay testing at Month 0 (V1;before dose 1)and at 1 month after dose 2(V5 for G1,V10 for G2:window 28-42 days);at least 1 determinate MenA/C/W/Y or MenB assay result at V5 and V10;received no prohibited treatment and had no protocol deviations through V5(G1)or V10(G2).
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1 (MenABCWY 0- and 12-Month Schedule)
Number analyzed (Participants) | 116
Percentage of participants
  A22: number analyzed (Participants) | 114
  A22 | 7.0 [3.1 to 13.4]
  A56 | 2.6 [0.5 to 7.4]
  B24 | 1.7 [0.2 to 6.1]
  B44 | 0.9 [0.0 to 4.7]

2. Primary Outcome: Percentage of Participants With hSBA Titer >=LLOQ for Each of the 4 Primary MenB Test Strains at 1 Month After Vaccination 2: 0 and 12 Month Schedule
Description: Percentage of participants achieving hSBA titer >=LLOQ (1:16 for strain A22 and 1:8 for strains A56, B24, and B44) for each of the 4 primary MenB test strains at 1 month after vaccination 2 in participants who received MenABCWY at Month 0 and Month 12 were reported in this outcome measure. "Number analyzed" = number of participants evaluable at specific rows.
Time Frame: 1 month after vaccination 2 (second dose of MenABCWY)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1 (MenABCWY 0- and 12-Month Schedule)
Number analyzed (Participants) | 116
Percentage of participants
  A22: number analyzed (Participants) | 113
  A22 | 99.1 [95.2 to 100.0]
  A56: number analyzed (Participants) | 115
  A56 | 100.0 [96.8 to 100.0]
  B24: number analyzed (Participants) | 113
  B24 | 98.2 [93.8 to 99.8]
  B44 | 96.6 [91.4 to 99.1]

3. Primary Outcome: Percentage of Participants With hSBA Titer >= LLOQ for Each of the 4 Primary MenB Test Strains at Baseline: 0 and 36 Month Schedule
Description: Percentage of participants achieving hSBA titer >=LLOQ (1:16 for strain A22 and 1:8 for strains A56, B24, and B44) for each of the 4 primary MenB test strains at baseline were reported in this outcome measure. "Number of Participants Analyzed"= number of participants evaluable for this outcome measure and "Number analyzed" = number of participants evaluable at specific rows.
Time Frame: Baseline (before vaccination 1)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 2 (MenABCWY 0- and 36-Month Schedule)
Number analyzed (Participants) | 99
Percentage of participants
  A22: number analyzed (Participants) | 90
  A22 | 10.0 [4.7 to 18.1]
  A56: number analyzed (Participants) | 95
  A56 | 1.1 [0.0 to 5.7]
  B24 | 2.0 [0.2 to 7.1]
  B44 | 1.0 [0.0 to 5.5]

4. Primary Outcome: Percentage of Participants With hSBA Titer >= LLOQ for Each of the 4 Primary MenB Test Strains at 1 Month After Vaccination 3: 0 and 36 Month Schedule
Description: Percentage of participants achieving hSBA titer >=LLOQ (1:16 for strain A22 and 1:8 for strains A56, B24, and B44) for each of the 4 primary MenB test strains at 1 month after vaccination 3 (second dose of MenABCWY) in participants who received MenABCWY at Month 0 and Month 36. "Number of Participants Analyzed"= number of participants evaluable for this outcome measure and "Number analyzed" = number of participants evaluable at specific rows.
Time Frame: 1 Month After Vaccination 3 (second dose of MenABCWY)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 2 (MenABCWY 0- and 36-Month Schedule)
Number analyzed (Participants) | 99
Percentage of participants
  A22 | 100.0 [96.3 to 100.0]
  A56: number analyzed (Participants) | 96
  A56 | 100.0 [96.2 to 100.0]
  B24 | 100.0 [96.3 to 100.0]
  B44: number analyzed (Participants) | 98
  B44 | 100.0 [96.3 to 100.0]

5. Primary Outcome: Percentage of Participants Reporting Adverse Events (AEs) Within 30 Days After Vaccination 1: 0 and 12 Month Schedule
Description: An AE was defined as any untoward medical occurrence in a participant, temporally associated with the use of investigational product, whether or not considered related to the investigational product. AEs included both serious and all non-serious adverse events.
Time Frame: Within 30 days after vaccination 1 (first dose of MenABCWY)
Population: Vaccination 1 safety population included participants who received the first dose of study intervention at Visit 1 and for whom safety information from Visit 1 up to Visit 4 was available in Groups 1 and 2.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1 (MenABCWY 0- and 12-Month Schedule)
Number analyzed (Participants) | 146
Percentage of participants | 28.8 [21.6 to 36.8]

6. Primary Outcome: Percentage of Participants Reporting AEs Within 30 Days After Vaccination 2: 0 and 12 Month Schedule
Description: An AE was any untoward medical occurrence in a participant, temporally associated with the use of investigational product, whether or not considered related to the investigational product. AEs included both serious and all non-serious adverse events.
Time Frame: Within 30 days after vaccination 2 (second dose of MenABCWY)
Population: Vaccination 2 safety population included participants who received the second dose of study intervention at Visit 4 (MenABCWY for Group 1, saline for Group 2) and for whom safety information from Visit 4 up to Visit 7 (for Group 1) or Visit 9 (for Group 2) was available.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1 (MenABCWY 0- and 12-Month Schedule)
Number analyzed (Participants) | 121
Percentage of participants | 15.7 [9.7 to 23.4]

7. Primary Outcome: Percentage of Participants Reporting AEs Within 30 Days After Vaccination 1: 0 and 36 Month Schedule
Description: as for outcome 6
Time Frame: Within 30 days after vaccination 1 (first dose of MenABCWY)
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 2 (MenABCWY 0- and 36-Month Schedule)
Number analyzed (Participants) | 148
Percentage of participants | 27.7 [20.7 to 35.7]

8. Primary Outcome: Percentage of Participants Reporting AEs Within 30 Days After Vaccination 2: 0 and 36 Month Schedule
Description: as for outcome 6
Time Frame: Within 30 days after vaccination 2 (saline)
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 2 (MenABCWY 0- and 36-Month Schedule)
Number analyzed (Participants) | 130
Percentage of participants | 13.8 [8.4 to 21.0]

9. Primary Outcome: Percentage of Participants Reporting AEs Within 30 Days After Vaccination 3: 0 and 36 Month Schedule
Description: as for outcome 6
Time Frame: Within 30 days after vaccination 3 (second dose of MenABCWY)
Population: Vaccination 3 safety population included participants who received the third dose of study intervention at Visit 9 (MenABCWY for Group 2) and for whom safety information from Visit 9 through Visit 10 was available.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 2 (MenABCWY 0- and 36-Month Schedule)
Number analyzed (Participants) | 103
Percentage of participants | 19.4 [12.3 to 28.4]

10. Primary Outcome: Percentage of Participants Reporting Serious Adverse Events (SAEs), Medically Attended Adverse Events (MAEs) and Newly Diagnosed Chronic Medical Condition (NDCMCs) Within 30 Days After Vaccination 1: 0 and 12 Month Schedule
Description: An AE was any untoward medical occurrence in a participant, temporally associated with the use of investigational product, whether or not considered related to the investigational product. An SAE was any untoward medical occurrence that, at any dose: resulted in death; required inpatient hospitalization or prolongation of existing hospitalization; was life threatening; resulted in persistent disability/incapacity; congenital anomaly/birth defect and other important medical events. An MAE was defined as a non-serious AE (other than serious AE) that resulted in an evaluation at a medical facility. An NDCMC was defined as a disease or medical condition, not previously identified, that was expected to be persistent or otherwise long-lasting in its effects.
Time Frame: Within 30 days after vaccination 1 (First dose of MenABCWY)
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1 (MenABCWY 0- and 12-Month Schedule)
Number analyzed (Participants) | 146
Percentage of participants
  SAEs | 0.0 [0.0 to 2.5]
  MAEs | 6.2 [2.9 to 11.4]
  NDCMCs | 0.7 [0.0 to 3.8]

11. Primary Outcome: Percentage of Participants Reporting SAEs, MAEs and NDCMCs Within 30 Days After Vaccination 2: 0 and 12 Month Schedule
Description: An AE was any untoward medical occurrence in a participant, temporally associated with the use of investigational product, whether or not considered related to the investigational product. An SAE was any untoward medical occurrence that, at any dose: resulted in death; required inpatient hospitalization or prolongation of existing hospitalization; was life threatening; resulted in persistent disability/incapacity; congenital anomaly/birth defect and other important medical events. An MAE was defined as a nonserious AE that resulted in an evaluation at a medical facility. An NDCMC was defined as a disease or medical condition, not previously identified, that was expected to be persistent or otherwise long-lasting in its effects.
Time Frame: Within 30 days after vaccination 2 (Second dose of MenABCWY)
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1 (MenABCWY 0- and 12-Month Schedule)
Number analyzed (Participants) | 121
Percentage of participants
  SAEs | 0.0 [0.0 to 3.0]
  MAEs | 5.0 [1.8 to 10.5]
  NDCMCs | 0.0 [0.0 to 3.0]

12. Primary Outcome: Percentage of Participants Reporting SAEs, MAEs and NDCMCs Within 30 Days After Vaccination 1: 0 and 36 Month Schedule
Description: as for outcome 11
Time Frame: Within 30 days after vaccination 1 (First dose of MenABCWY)
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 2 (MenABCWY 0- and 36-Month Schedule)
Number analyzed (Participants) | 148
Percentage of participants
  SAEs | 0.0 [0.0 to 2.5]
  MAEs | 7.4 [3.8 to 12.9]
  NDCMCs | 0.0 [0.0 to 2.5]

13. Primary Outcome: Percentage of Participants Reporting SAEs, MAEs and NDCMCs Within 30 Days After Vaccination 2: 0 and 36 Month Schedule
Description: as for outcome 11
Time Frame: Within 30 days after vaccination 2 (Saline)
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 2 (MenABCWY 0- and 36-Month Schedule)
Number analyzed (Participants) | 130
Percentage of participants
  SAEs | 0.0 [0.0 to 2.8]
  MAEs | 6.9 [3.2 to 12.7]
  NDCMCs | 0.8 [0.0 to 4.2]

14. Primary Outcome: Percentage of Participants Reporting SAEs, MAEs and NDCMCs Within 30 Days After Vaccination 3: 0 and 36 Month Schedule
Description: as for outcome 11
Time Frame: Within 30 days after vaccination 3 (Second dose of MenABCWY)
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 2 (MenABCWY 0- and 36-Month Schedule)
Number analyzed (Participants) | 103
Percentage of participants
  SAEs | 0.0 [0.0 to 3.5]
  MAEs | 1.9 [0.2 to 6.8]
  NDCMCs | 0.0 [0.0 to 3.5]

15. Primary Outcome: Percentage of Participants Reporting AEs Within 30 Days After Any MenABCWY Vaccination: 0 and 12 Month Schedule
Description: as for outcome 6
Time Frame: Within 30 Days after any MenABCWY vaccination
Population: Safety population set included all randomized participants who received at least 1 dose of the study intervention and had safety data reported after vaccination.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1 (MenABCWY 0- and 12-Month Schedule)
Number analyzed (Participants) | 146
Percentage of participants | 34.9 [27.2 to 43.3]

16. Primary Outcome: Percentage of Participants Reporting AEs Within 30 Days After Any MenABCWY Vaccination: 0 and 36 Month Schedule
Description: as for outcome 6
Time Frame: Within 30 days after any MenABCWY vaccination
Population: as for outcome 15
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 2 (MenABCWY 0- and 36-Month Schedule)
Number analyzed (Participants) | 148
Percentage of participants | 32.4 [25.0 to 40.6]

17. Primary Outcome: Percentage of Participants Reporting SAEs, MAEs and NDCMCs Within 30 Days After Any MenABCWY Vaccination: 0 and 12 Month Schedule
Description: as for outcome 11
Time Frame: Within 30 days after any MenABCWY vaccination
Population: as for outcome 15
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1 (MenABCWY 0- and 12-Month Schedule)
Number analyzed (Participants) | 146
Percentage of participants
  SAEs | 0.0 [0.0 to 2.5]
  MAEs | 10.3 [5.9 to 16.4]
  NDCMCs | 0.7 [0.0 to 3.8]

18. Primary Outcome: Percentage of Participants Reporting SAEs, MAEs and NDCMCs Within 30 Days After Any MenABCWY Vaccination: 0 and 36 Month Schedule
Description: as for outcome 11
Time Frame: Within 30 days after any MenABCWY vaccination
Population: as for outcome 15
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 2 (MenABCWY 0- and 36-Month Schedule)
Number analyzed (Participants) | 148
Percentage of participants
  SAEs | 0.0 [0.0 to 2.5]
  MAEs | 8.8 [4.8 to 14.6]
  NDCMCs | 0.0 [0.0 to 2.5]

19. Primary Outcome: Percentage of Participants Reporting AEs From Vaccination 1 Through 1 Month After Vaccination 1: 0 and 12 Month Schedule
Description: as for outcome 6
Time Frame: From vaccination 1 through 1 month after vaccination 1 (First dose of MenABCWY)
Population: Vaccination 1 safety population included all participants who received the first dose of study intervention at Visit 1 and for whom safety information from Visit 1 up to Visit 4 was available in Groups 1 and 2.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1 (MenABCWY 0- and 12-Month Schedule)
Number analyzed (Participants) | 146
Percentage of participants | 30.8 [23.5 to 39.0]

20. Primary Outcome: Percentage of Participants Reporting AEs From Vaccination 1 Through 1 Month After Vaccination 1: 0 and 36 Month Schedule
Description: as for outcome 6
Time Frame: Vaccination 1 through 1 month after vaccination 1 (First dose of MenABCWY)
Population: as for outcome 19
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 2 (MenABCWY 0- and 36-Month Schedule)
Number analyzed (Participants) | 148
Percentage of participants | 29.1 [21.9 to 37.1]

21. Primary Outcome: Percentage of Participants Reporting SAEs, MAEs and NDCMCs From Vaccination 1 Through 1 Month After Vaccination 1: 0 and 12 Month Schedule
Description: as for outcome 11
Time Frame: From vaccination 1 through 1 month after vaccination 1 (First dose of MenABCWY)
Population: as for outcome 19
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1 (MenABCWY 0- and 12-Month Schedule)
Number analyzed (Participants) | 146
Percentage of participants
  SAEs | 0.0 [0.0 to 2.5]
  MAEs | 8.2 [4.3 to 13.9]
  NDCMCs | 0.7 [0.0 to 3.8]

22. Primary Outcome: Percentage of Participants Reporting SAEs, MAEs and NDCMCs From Vaccination 1 Through 1 Month After Vaccination 1: 0 and 36 Month Schedule
Description: as for outcome 11
Time Frame: From vaccination 1 through 1 month after vaccination 1 (First dose of MenABCWY)
Population: as for outcome 19
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 2 (MenABCWY 0- and 36-Month Schedule)
Number analyzed (Participants) | 148
Percentage of participants
  SAEs | 0.0 [0.0 to 2.5]
  MAEs | 8.8 [4.8 to 14.6]
  NDCMCs | 0.0 [0.0 to 2.5]

23. Primary Outcome: Percentage of Participants Reporting AEs From Vaccination 2 Through 1 Month After Vaccination 2: 0 and 12 Month Schedule
Description: as for outcome 6
Time Frame: From vaccination 2 through 1 month after vaccination 2 (Second dose of MenABCWY)
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1 (MenABCWY 0- and 12-Month Schedule)
Number analyzed (Participants) | 121
Percentage of participants | 15.7 [9.7 to 23.4]

24. Primary Outcome: Percentage of Participants Reporting AEs From Vaccination 2 Through 1 Month After Vaccination 2: 0 and 36 Month Schedule
Description: as for outcome 6
Time Frame: From vaccination 2 through 1 month after vaccination 2 (Saline)
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 2 (MenABCWY 0- and 36-Month Schedule)
Number analyzed (Participants) | 130
Percentage of participants | 16.2 [10.3 to 23.6]

25. Primary Outcome: Percentage of Participants Reporting SAEs, MAEs and NDCMCs From Vaccination 2 Through 1 Month After Vaccination 2: 0 and 12 Month Schedule
Description: as for outcome 11
Time Frame: From vaccination 2 through 1 month after vaccination 2 (Second dose of MenABCWY)
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1 (MenABCWY 0- and 12-Month Schedule)
Number analyzed (Participants) | 121
Percentage of participants
  SAEs | 0.0 [0.0 to 3.0]
  MAEs | 5.0 [1.8 to 10.5]
  NDCMCs | 0.0 [0.0 to 3.0]

26. Primary Outcome: Percentage of Participants Reporting SAEs, MAEs and NDCMCs From Vaccination 2 Through 1 Month After Vaccination 2: 0 and 36 Month Schedule
Description: as for outcome 11
Time Frame: From vaccination 2 through 1 month after vaccination 2 (Saline)
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 2 (MenABCWY 0- and 36-Month Schedule)
Number analyzed (Participants) | 130
Percentage of participants
  SAEs | 0.0 [0.0 to 2.8]
  MAEs | 6.9 [3.2 to 12.7]
  NDCMCs | 1.5 [0.2 to 5.4]

27. Primary Outcome: Percentage of Participants Reporting AEs From Vaccination 3 Through 1 Month After Vaccination 3: 0 and 36 Month Schedule
Description: as for outcome 6
Time Frame: From vaccination 3 through 1 month after vaccination 3 (Second dose of MenABCWY)
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 2 (MenABCWY 0- and 36-Month Schedule)
Number analyzed (Participants) | 103
Percentage of participants | 19.4 [12.3 to 28.4]

28. Primary Outcome: Percentage of Participants Reporting SAEs, MAEs and NDCMCs From Vaccination 3 Through 1 Month After Vaccination 3: 0 and 36 Month Schedule
Description: as for outcome 11
Time Frame: From vaccination 3 through 1 month after vaccination 3 (Second dose of MenABCWY)
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 2 (MenABCWY 0- and 36-Month Schedule)
Number analyzed (Participants) | 103
Percentage of participants
  SAEs | 0.0 [0.0 to 3.5]
  MAEs | 3.9 [1.1 to 9.6]
  NDCMCs | 0.0 [0.0 to 3.5]

29. Primary Outcome: Percentage of Participants Reporting SAEs, MAEs and NDCMCs From 1 Month After Vaccination 1 Through 6 Months After Vaccination 1: 0 and 12 Month Schedule
Description: as for outcome 11
Time Frame: From 1 month after vaccination 1 through 6 months after vaccination 1 (First dose of MenABCWY)
Population: Follow-up safety population 1 included participants who received the first dose of study intervention and for whom safety information from Visit 2 up to Visit 4 in Groups 1 and 2 was available.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1 (MenABCWY 0- and 12-Month Schedule)
Number analyzed (Participants) | 145
Percentage of participants
  SAEs | 0.7 [0.0 to 3.8]
  MAEs | 16.6 [10.9 to 23.6]
  NDCMCs | 0.7 [0.0 to 3.8]

30. Primary Outcome: Percentage of Participants Reporting SAEs, MAEs and NDCMCs From 1 Month After Vaccination 1 Through 6 Months After Vaccination 1: 0 and 36 Month Schedule
Description: as for outcome 11
Time Frame: From 1 month after vaccination 1 through 6 months after vaccination 1 (First dose of MenABCWY)
Population: as for outcome 29
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 2 (MenABCWY 0- and 36-Month Schedule)
Number analyzed (Participants) | 148
Percentage of participants
  SAEs | 0.0 [0.0 to 2.5]
  MAEs | 14.2 [9.0 to 20.9]
  NDCMCs | 0.7 [0.0 to 3.7]

31. Primary Outcome: Percentage of Participants Reporting SAEs, MAEs and NDCMCs From 1 Month After Vaccination 2 Through 6 Months After Vaccination 2: 0 and 12 Month Schedule
Description: as for outcome 11
Time Frame: From 1 month after vaccination 2 through 6 months after vaccination 2 (Second dose of MenABCWY)
Population: Follow-up safety population 2 included participants who received the second dose of study intervention (MenABCWY for Group 1, saline for Group 2) and for whom safety information from Visit 5 up to Visit 7 (for Group 1) or Visit 9 (for Group 2) was available. Here, 'Number of Participants Analyzed' signifies participants evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1 (MenABCWY 0- and 12-Month Schedule)
Number analyzed (Participants) | 118
Percentage of participants
  SAEs | 0.8 [0.0 to 4.6]
  MAEs | 8.5 [4.1 to 15.0]
  NDCMCs | 0.0 [0.0 to 3.1]

32. Primary Outcome: Percentage of Participants Reporting SAEs, MAEs and NDCMCs From 1 Month After Vaccination 2 Through 6 Months After Vaccination 2: 0 and 36 Month Schedule
Description: as for outcome 11
Time Frame: From 1 month after vaccination 2 through 6 months after vaccination 2 (Saline)
Population: as for outcome 31
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 2 (MenABCWY 0- and 36-Month Schedule)
Number analyzed (Participants) | 128
Percentage of participants
  SAEs | 1.6 [0.2 to 5.5]
  MAEs | 9.4 [4.9 to 15.8]
  NDCMCs | 3.1 [0.9 to 7.8]

33. Primary Outcome: Percentage of Participants Reporting SAEs, MAEs and NDCMCs From Vaccination 1 Through 6 Months After Vaccination 1: 0 and 12 Month Schedule
Description: as for outcome 11
Time Frame: From vaccination 1 through 6 months after vaccination 1 (First dose of MenABCWY)
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1 (MenABCWY 0- and 12-Month Schedule)
Number analyzed (Participants) | 146
Percentage of participants
  SAEs | 0.7 [0.0 to 3.8]
  MAEs | 23.3 [16.7 to 31.0]
  NDCMCs | 1.4 [0.2 to 4.9]

34. Primary Outcome: Percentage of Participants Reporting SAEs, MAEs and NDCMCs From Vaccination 1 Through 6 Months After Vaccination 1: 0 and 36 Month Schedule
Description: as for outcome 11
Time Frame: From vaccination 1 through 6 months after vaccination 1 (First dose of MenABCWY)
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 2 (MenABCWY 0- and 36-Month Schedule)
Number analyzed (Participants) | 148
Percentage of participants
  SAEs | 0.0 [0.0 to 2.5]
  MAEs | 19.6 [13.5 to 26.9]
  NDCMCs | 0.7 [0.0 to 3.7]

35. Primary Outcome: Percentage of Participants Reporting SAEs, MAEs and NDCMCs From Vaccination 2 Through 6 Months After Vaccination 2: 0 and 12 Month Schedule
Description: as for outcome 11
Time Frame: From vaccination 2 through 6 months after vaccination 2 (Second dose of MenABCWY)
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1 (MenABCWY 0- and 12-Month Schedule)
Number analyzed (Participants) | 121
Percentage of participants
  SAEs | 0.8 [0.0 to 4.5]
  MAEs | 13.2 [7.8 to 20.6]
  NDCMCs | 0.0 [0.0 to 3.0]

36. Primary Outcome: Percentage of Participants Reporting SAEs, MAEs and NDCMCs From Vaccination 2 Through 6 Months After Vaccination 2: 0 and 36 Month Schedule
Description: as for outcome 11
Time Frame: From vaccination 2 through 6 months after vaccination 2 (Saline)
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 2 (MenABCWY 0- and 36-Month Schedule)
Number analyzed (Participants) | 130
Percentage of participants
  SAEs | 1.5 [0.2 to 5.4]
  MAEs | 14.6 [9.0 to 21.9]
  NDCMCs | 4.6 [1.7 to 9.8]

37. Primary Outcome: Percentage of Participants Reporting at Least 1 Immediate AE After Vaccination 1: 0 and 12 Month Schedule
Description: Immediate AEs were defined as AEs occurring within the first 30 minutes after study intervention administration.
Time Frame: 30 minutes after vaccination 1 (First dose of MenABCWY)
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1 (MenABCWY 0- and 12-Month Schedule)
Number analyzed (Participants) | 146
Percentage of participants | 0.7 [0.0 to 3.8]

38. Primary Outcome: Percentage of Participants Reporting at Least 1 Immediate AE After Vaccination 2: 0 and 12 Month Schedule
Description: Immediate AEs were defined as AEs occurring within the first 30 minutes after study intervention administration.
Time Frame: 30 minutes after vaccination 2 (Second dose of MenABCWY)
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1 (MenABCWY 0- and 12-Month Schedule)
Number analyzed (Participants) | 121
Percentage of participants | 0.0 [0.0 to 3.0]

39. Primary Outcome: Percentage of Participants Reporting at Least 1 Immediate AE After Vaccination 1: 0 and 36 Month Schedule
Description: Immediate AEs were defined as AEs occurring within the first 30 minutes after study intervention administration.
Time Frame: 30 minutes after vaccination 1 (First dose of MenABCWY)
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 2 (MenABCWY 0- and 36-Month Schedule)
Number analyzed (Participants) | 148
Percentage of participants | 0.7 [0.0 to 3.7]

40. Primary Outcome: Percentage of Participants Reporting at Least 1 Immediate AE After Vaccination 2: 0 and 36 Month Schedule
Description: Immediate AEs were defined as AEs occurring within the first 30 minutes after study intervention administration.
Time Frame: 30 minutes after vaccination 2 (Saline)
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 2 (MenABCWY 0- and 36-Month Schedule)
Number analyzed (Participants) | 130
Percentage of participants | 1.5 [0.2 to 5.4]

41. Primary Outcome: Percentage of Participants Reporting at Least 1 Immediate AE After Vaccination 3: 0 and 36 Month Schedule
Description: Immediate AEs were defined as AEs occurring within the first 30 minutes after study intervention administration.
Time Frame: 30 minutes after vaccination 3 (Second dose of MenABCWY)
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 2 (MenABCWY 0- and 36-Month Schedule)
Number analyzed (Participants) | 103
Percentage of participants | 2.9 [0.6 to 8.3]

42. Primary Outcome: Percentage of Participants Who Missed School or Work Because of AEs Within 6 Months After Vaccination 1: 0 and 12 Month Schedule
Description: An AE was any untoward medical occurrence in a participant, temporally associated with the use of investigational product, whether or not considered related to the investigational product.
Time Frame: Within 6 months after vaccination 1 (First dose of MenABCWY)
Population: as for outcome 5
Measure: Number; unit: Percentage of participants
Arm/Group | Group 1 (MenABCWY 0- and 12-Month Schedule)
Number analyzed (Participants) | 146
Percentage of participants | 8.2

43. Primary Outcome: Percentage of Participants Who Missed School or Work Because of AEs Within 6 Months After Vaccination 1: 0 and 36 Month Schedule
Description: as for outcome 42
Time Frame: Within 6 months after vaccination 1 (First dose of MenABCWY)
Population: as for outcome 5
Measure: Number; unit: Percentage of participants
Arm/Group | Group 2 (MenABCWY 0- and 36-Month Schedule)
Number analyzed (Participants) | 148
Percentage of participants | 8.1

44. Primary Outcome: Percentage of Participants Who Missed School or Work Because of AEs Within 6 Months After Vaccination 2: 0 and 12 Month Schedule
Description: as for outcome 42
Time Frame: Within 6 months after vaccination 2 (Second dose of MenABCWY)
Population: as for outcome 6
Measure: Number; unit: Percentage of participants
Arm/Group | Group 1 (MenABCWY 0- and 12-Month Schedule)
Number analyzed (Participants) | 121
Percentage of participants | 8.3

45. Primary Outcome: Percentage of Participants Who Missed School or Work Because of AEs Within 6 Months After Vaccination 2: 0 and 36 Month Schedule
Description: as for outcome 42
Time Frame: Within 6 months after vaccination 2 (Saline)
Population: as for outcome 6
Measure: Number; unit: Percentage of participants
Arm/Group | Group 2 (MenABCWY 0- and 36-Month Schedule)
Number analyzed (Participants) | 130
Percentage of participants | 6.2

46. Primary Outcome: Percentage of Participants Who Missed School or Work Because of AEs Within 1 Month After Vaccination 3: 0 and 36 Month Schedule
Description: as for outcome 42
Time Frame: Within 1 month after vaccination 3 (Second dose of MenABCWY)
Population: as for outcome 9
Measure: Number; unit: Percentage of participants
Arm/Group | Group 2 (MenABCWY 0- and 36-Month Schedule)
Number analyzed (Participants) | 103
Percentage of participants | 1.9

47. Secondary Outcome: Percentage of Participants With hSBA Titer >= LLOQ for Each of the Meningococcal Group A, C, W, and Y (MenACWY) Test Strains at Baseline and 1 Month After the First Dose of MenABCWY: 0 and 12 Month Schedule-Post-Vaccination 1 Evaluable Population
Description: Percentage of participants achieving hSBA titer >=LLOQ (LLOQ = 1:8 for all MenA, MenC, MenW, and MenY serogroups) for each of the MenACWY test strains at baseline and one month after first dose of MenABCWY in participants who received the first dose of MenABCWY were reported in this outcome measure. "Number analyzed" = number of participants evaluable at specific rows.
Time Frame: Baseline (before vaccination 1) and 1 month after the first dose of MenABCWY
Population: PV1 EP: all randomized participants, eligible throughout Visit 2, received study intervention at Visit 1 as randomized, had blood drawn for assay testing within required time frames at Month 0 (Visit 1; before Vaccination 1) and Month 1 (Visit 2; 1 month after the first vaccination: window 28-42 days) had at least 1 valid and determinate MenA/C/W/Y assay result at Visit 2, had received no prohibited vaccines or treatment through Visit 2 and had no important protocol deviations through Visit 2.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1 (MenABCWY 0- and 12-Month Schedule)
Number analyzed (Participants) | 140
Percentage of participants
  MenA: Baseline | 10.7 [6.1 to 17.1]
  MenA: 1 month after the first dose of MenABCWY | 98.6 [94.9 to 99.8]
  MenC: Baseline: number analyzed (Participants) | 139
  MenC: Baseline | 10.1 [5.6 to 16.3]
  MenC: 1 month after the first dose of MenABCWY | 79.3 [71.6 to 85.7]
  MenW: Baseline: number analyzed (Participants) | 138
  MenW: Baseline | 15.9 [10.3 to 23.1]
  MenW: 1 month after the first dose of MenABCWY | 98.6 [94.9 to 99.8]
  MenY: Baseline: number analyzed (Participants) | 136
  MenY: Baseline | 36.0 [28.0 to 44.7]
  MenY: 1 month after the first dose of MenABCWY | 99.3 [96.1 to 100.0]

48. Secondary Outcome: Percentage of Participants With hSBA Titer >= LLOQ for Each of the MenACWY Test Strains at Baseline and 1 Month After the Second Dose of MenABCWY: 0 and 12 Month Schedule-Post-Vaccination 2 Evaluable Population
Description: Percentage of participants achieving hSBA titer >=LLOQ (LLOQ = 1:8 for all MenA, MenC, MenW, and MenY serogroups) for each of the MenACWY test strains at baseline and one month after second dose of MenABCWY in participants who received the first and second dose of MenABCWY were reported in this outcome measure. "Number analyzed" = number of participants evaluable at specific rows.
Time Frame: Baseline (before vaccination 1) and 1 month after the second dose of MenABCWY
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1 (MenABCWY 0- and 12-Month Schedule)
Number analyzed (Participants) | 116
Percentage of participants
  MenA: Baseline | 6.9 [3.0 to 13.1]
  MenA: 1 month after the second dose of MenABCWY | 99.1 [95.3 to 100.0]
  MenC: Baseline: number analyzed (Participants) | 115
  MenC: Baseline | 9.6 [4.9 to 16.5]
  MenC: 1 month after the second dose of MenABCWY | 99.1 [95.3 to 100.0]
  MenW: Baseline: number analyzed (Participants) | 114
  MenW: Baseline | 16.7 [10.3 to 24.8]
  MenW: 1 month after the second dose of MenABCWY: number analyzed (Participants) | 115
  MenW: 1 month after the second dose of MenABCWY | 100.0 [96.8 to 100.0]
  MenY: Baseline: number analyzed (Participants) | 113
  MenY: Baseline | 32.7 [24.2 to 42.2]
  MenY: 1 month after the second dose of MenABCWY: number analyzed (Participants) | 114
  MenY: 1 month after the second dose of MenABCWY | 100.0 [96.8 to 100.0]

49. Secondary Outcome: Percentage of Participants With hSBA Titer >=LLOQ for Each of the MenACWY Test Strains at Baseline and 1 Month After First Dose of MenABCWY: 0 and 36 Month Schedule-Post-Vaccination 1 Evaluable Population
Description: Percentage of participants achieving hSBA titer >=LLOQ (LLOQ = 1:8 for all MenA, MenC, MenW, and MenY serogroups) for each of the MenACWY test strains at baseline and one month after first dose of MenABCWY in participants who received who received the first dose of MenABCWY were reported in this outcome measure. "Number analyzed" = number of participants evaluable at specific rows.
Time Frame: Baseline (before vaccination 1) and 1 month after first dose of MenABCWY
Population: as for outcome 47
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 2 (MenABCWY 0- and 36-Month Schedule)
Number analyzed (Participants) | 144
Percentage of participants
  MenA: Baseline: number analyzed (Participants) | 141
  MenA: Baseline | 7.1 [3.5 to 12.7]
  MenA: 1 month after the first dose of MenABCWY | 100.0 [97.5 to 100.0]
  MenC: Baseline | 10.4 [5.9 to 16.6]
  MenC: 1 month after the first dose of MenABCWY: number analyzed (Participants) | 143
  MenC: 1 month after the first dose of MenABCWY | 80.4 [73.0 to 86.6]
  MenW: Baseline: number analyzed (Participants) | 143
  MenW: Baseline | 15.4 [9.9 to 22.4]
  MenW: 1 month after the first dose of MenABCWY | 98.6 [95.1 to 99.8]
  MenY: Baseline: number analyzed (Participants) | 142
  MenY: Baseline | 35.2 [27.4 to 43.7]
  MenY: 1 month after the first dose of MenABCWY: number analyzed (Participants) | 143
  MenY: 1 month after the first dose of MenABCWY | 99.3 [96.2 to 100.0]

50. Secondary Outcome: Percentage of Participants With hSBA Titer >=LLOQ for Each of the MenACWY Test Strains at Baseline and 1 Month After Second Dose of MenABCWY: 0 and 36 Month Schedule-Post-Vaccination 2 Evaluable Population
Description: Percentage of participants achieving hSBA titer >=LLOQ (LLOQ = 1:8 for all MenA, MenC, MenW, and MenY serogroups) for each of the meningococcal group A, C, W, and Y (MenACWY) test strains at baseline and one month after second dose of MenABCWY in participants who received the first and second dose of MenABCWY were reported in this outcome measure. "Number of Participants Analyzed"= number of participants evaluable for this outcome measure and "Number analyzed" = number of participants evaluable at specific rows.
Time Frame: Baseline (before vaccination 1) and 1 month after second dose of MenABCWY
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 2 (MenABCWY 0- and 36-Month Schedule)
Number analyzed (Participants) | 100
Percentage of participants
  MenA: Baseline: number analyzed (Participants) | 99
  MenA: Baseline | 7.1 [2.9 to 14.0]
  MenA: 1 month after the second dose of MenABCWY: number analyzed (Participants) | 95
  MenA: 1 month after the second dose of MenABCWY | 100.0 [96.2 to 100.0]
  MenC: Baseline | 12.0 [6.4 to 20.0]
  MenC: 1 month after the second dose of MenABCWY: number analyzed (Participants) | 83
  MenC: 1 month after the second dose of MenABCWY | 100.0 [95.7 to 100.0]
  MenW: Baseline: number analyzed (Participants) | 99
  MenW: Baseline | 16.2 [9.5 to 24.9]
  MenW: 1 month after the second dose of MenABCWY: number analyzed (Participants) | 89
  MenW: 1 month after the second dose of MenABCWY | 100.0 [95.9 to 100.0]
  MenY: Baseline: number analyzed (Participants) | 98
  MenY: Baseline | 37.8 [28.2 to 48.1]
  MenY: 1 month after the second dose of MenABCWY: number analyzed (Participants) | 89
  MenY: 1 month after the second dose of MenABCWY | 100.0 [95.9 to 100.0]

51. Secondary Outcome: Percentage of Participants With hSBA Titer >=LLOQ for Each of the 4 Primary MenB Test Strains at 12 Months and 24 Months After Vaccination 2: 0 and 12 Month Schedule
Description: Percentage of participants achieving hSBA titer >=LLOQ for each of the 4 primary MenB test strains (1:16 for strain A22 and 1:8 for strains A56, B24, and B44) at 12 and 24 months after the second dose of MenABCWY were reported in this outcome measure. "Number of Participants Analyzed"= number of participants evaluable for this outcome measure and "Number analyzed" = number of participants evaluable at specific rows.
Time Frame: At 12 months and 24 months after vaccination 2 (Second dose of MenABCWY)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1 (MenABCWY 0- and 12-Month Schedule)
Number analyzed (Participants) | 110
Percentage of participants
  A22: At 12 months: number analyzed (Participants) | 109
  A22: At 12 months | 79.8 [71.1 to 86.9]
  A56: At 12 months: number analyzed (Participants) | 107
  A56: At 12 months | 86.0 [77.9 to 91.9]
  B24: At 12 months: number analyzed (Participants) | 107
  B24: At 12 months | 43.0 [33.5 to 52.9]
  B44: At 12 months | 55.5 [45.7 to 64.9]
  A22: At 24 months: number analyzed (Participants) | 98
  A22: At 24 months | 73.5 [63.6 to 81.9]
  A56: At 24 months: number analyzed (Participants) | 92
  A56: At 24 months | 75.0 [64.9 to 83.4]
  B24: At 24 months: number analyzed (Participants) | 100
  B24: At 24 months | 44.0 [34.1 to 54.3]
  B44: At 24 months: number analyzed (Participants) | 101
  B44: At 24 months | 50.5 [40.4 to 60.6]

52. Secondary Outcome: Percentage of Participants With hSBA Titer >=LLOQ for Each ACWY Test Strains at 12 Months and 24 Months After Vaccination 2: 0 and 12 Month Schedule
Description: Percentage of participants achieving hSBA titer >=LLOQ (LLOQ = 1:8 for all MenA, MenC, MenW, and MenY serogroups) for each of the ACWY test (MenA, MenC, MenW, MenY) at 12 and 24 months after the second dose of MenABCWY2 were reported in this outcome measure. "Number of Participants Analyzed"= number of participants evaluable for this outcome measure and "Number analyzed" = number of participants evaluable at specific rows.
Time Frame: At 12 months and 24 months after vaccination 2 (Second dose of MenABCWY)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1 (MenABCWY 0- and 12-Month Schedule)
Number analyzed (Participants) | 111
Percentage of participants
  MenA: At 12 months | 100.0 [96.7 to 100.0]
  MenC: At 12 months: number analyzed (Participants) | 107
  MenC: At 12 months | 93.5 [87.0 to 97.3]
  MenW: At 12 months: number analyzed (Participants) | 105
  MenW: At 12 months | 100.0 [96.5 to 100.0]
  MenY: At 12 months: number analyzed (Participants) | 104
  MenY: At 12 months | 99.0 [94.8 to 100.0]
  MenA: At 24 months: number analyzed (Participants) | 100
  MenA: At 24 months | 98.0 [93.0 to 99.8]
  MenC: At 24 months: number analyzed (Participants) | 99
  MenC: At 24 months | 88.9 [81.0 to 94.3]
  MenW: At 24 months: number analyzed (Participants) | 99
  MenW: At 24 months | 100.0 [96.3 to 100.0]
  MenY: At 24 months: number analyzed (Participants) | 97
  MenY: At 24 months | 100.0 [96.3 to 100.0]

ADVERSE EVENTS:
Time Frame: Group 1: Up to 36 months; Group 2: Up to 37 months
Description: Same event may appear as both an adverse event (AE) and serious adverse event (SAE). However, what is presented are distinct events. An event may be categorized as serious in 1 participant and as non-serious in another, or a participant may have experienced both a serious and non-serious event. Safety population set included all randomized participants who received at least 1 dose of the study intervention and had safety data reported after vaccination.
Arm/Group | Group 1 (MenABCWY 0- and 12-Month Schedule) | Group 2 (MenABCWY 0- and 36-Month Schedule)
All-Cause Mortality (participants affected / at risk) | 0/146 | 0/148
Serious Adverse Events (participants affected / at risk) | 2/146 | 2/148
Other Adverse Events (participants affected / at risk) | 64/146 | 64/148
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1 (MenABCWY 0- and 12-Month Schedule) (N=146) | Group 2 (MenABCWY 0- and 36-Month Schedule) (N=148)
Palpitations (Cardiac disorders) | 0 | 1
Chest pain (General disorders) | 0 | 1
Acute hepatic failure (Hepatobiliary disorders) | 1 | 0
Cellulitis orbital (Infections and infestations) | 1 | 0
Intentional overdose (Injury, poisoning and procedural complications) | 1 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1 (MenABCWY 0- and 12-Month Schedule) (N=146) | Group 2 (MenABCWY 0- and 36-Month Schedule) (N=148)
Injection site swelling (General disorders) | 0 | 4
Injection site warmth (General disorders) | 2 | 0
Pain (General disorders) | 2 | 9
Pyrexia (General disorders) | 11 | 8
Vaccination site erythema (General disorders) | 0 | 2
Vaccination site pain (General disorders) | 3 | 10
Diarrhoea (Gastrointestinal disorders) | 0 | 3
Nausea (Gastrointestinal disorders) | 2 | 4
Vomiting (Gastrointestinal disorders) | 6 | 6
COVID-19 (Infections and infestations) | 10 | 4
Gastroenteritis (Infections and infestations) | 0 | 2
Influenza (Infections and infestations) | 0 | 2
Nasopharyngitis (Infections and infestations) | 5 | 2
Pharyngitis (Infections and infestations) | 5 | 3
Pharyngitis streptococcal (Infections and infestations) | 1 | 2
Suspected COVID-19 (Infections and infestations) | 1 | 2
Upper respiratory tract infection (Infections and infestations) | 5 | 11
Fall (Injury, poisoning and procedural complications) | 4 | 5
Ligament sprain (Injury, poisoning and procedural complications) | 2 | 5
Limb injury (Injury, poisoning and procedural complications) | 3 | 3
Radius fracture (Injury, poisoning and procedural complications) | 1 | 2
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 2
Body temperature increased (Investigations) | 3 | 7
SARS-CoV-2 test positive (Investigations) | 0 | 2
Decreased appetite (Metabolism and nutrition disorders) | 1 | 2
Overweight (Metabolism and nutrition disorders) | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 2
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Dizziness (Nervous system disorders) | 1 | 2
Headache (Nervous system disorders) | 11 | 10
Attention deficit hyperactivity disorder (Psychiatric disorders) | 1 | 2
Depression (Psychiatric disorders) | 4 | 6
Generalised anxiety disorder (Psychiatric disorders) | 1 | 3
Insomnia (Psychiatric disorders) | 1 | 2
Suicidal ideation (Psychiatric disorders) | 1 | 2
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 2
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Cerumen impaction (Ear and labyrinth disorders) | 2 | 0
Chills (General disorders) | 3 | 1
Fatigue (General disorders) | 7 | 6
Injection site erythema (General disorders) | 5 | 5
Injection site pain (General disorders) | 15 | 15
Injection site rash (General disorders) | 2 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1 | 2
Abdominal Pain (Gastrointestinal disorders) | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publication until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2021-01-07): https://cdn.clinicaltrials.gov/large-docs/76/NCT04440176/Prot_000.pdf
  • Statistical Analysis Plan (2024-04-15): https://cdn.clinicaltrials.gov/large-docs/76/NCT04440176/SAP_001.pdf